CLINICAL TRIAL: NCT06338943
Title: Middle-aged Women With Adverse Pregnancy Outcomes and Heart Failure With Preserved Ejection Fraction
Acronym: MAPO-HF
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 02-02/24
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure Preserved Ejection Fraction; Pregnancy Complications
Keywords: Heart Failure Preserved Ejection Fraction; Adverse Pregnancy Outcomes; Arterial Hypertension; Gestational Diabetes; Mediation
MeSH Terms: conditions — Heart Failure, Diastolic; Pregnancy Complications; Hypertension; Diabetes, Gestational; Negotiating | interventions — Echocardiography; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with the history of pregnancy: Patient with the history of pregnancy (1 or more > 20 weeks)
  This group will further be subdivided in a subgroup with HFpEF and a group without HFpEF
  Interventions: Diagnostic Test: Echocardiography; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography to diagnose HFpEF
Other: Questionnaire — Questionnaire to determine the presence of adverse pregnancy outcomes history

SUMMARY:
Due to the steady increase in the burden of HFpEF, especially in women, it is an important task to search for new markers and early predictors associated with the development of this disease. Nowadays, the relationship of adverse pregnancy factors with the development of long-term cardiac pathology, in particular, HFpEF, has not been completely established. One of the most significant issue is studying the younger phenotype of women.

The goal of this observational analytical cross-sectional study is to study the relationship of heart failure with a preserved ejection fraction in middle-aged women with adverse pregnancy outcomes in the history of pregnancy.

Research question: is there an association between adverse pregnancy factors and the development of HF in middle-aged women?

Objectives

1. To assess the frequency of detection of APOs in the history of pregnancy in middle-aged women, depending on the presence or absence of HFpEF.
2. To compare clinical and anamnestic data, morphological and functional parameters of the heart in middle-aged women with the presence and absence of HFpEF.
3. To establish an association between APOs and the development of HFpEF in the long-term period in middle-aged women.
4. To identify mediators between the presence of APOs and the development of HFpEF in middle-aged women.

Study population - 45-60 year-old women with the history of pregnancy (>20 weeks) in the absence of low left ventricle ejection fraction (<50%)

Primary endpoint: The prevalence of HFpEF in patients with the history of APOs.

DETAILED DESCRIPTION:
Heart failure (HF) occupies a special place in the structure of cardiological pathology. This is largely due to the active modernization of approaches to the diagnosis of HF - every year the possibilities of cardiac imaging increase significantly, which leads to dynamic changes in the criteria for diagnosis. To the greatest extent, these changes affect heart failure with a preserved ejection fraction (HFpEF; left ventricular ejection fraction ≥ 50%), the importance of which is steadily growing with increasing life expectancy, obesity and cardiometabolic disorders. If in the recent past, HF was perceived not as independent disease, which is a complication of the underlying cardiac pathology, today, due to the increasing detectability of HFpEF, the latter can be considered as a separate multifactorial disease. Patients with HFpEF make up about half of the population of patients with HF, which, together with difficulties in understanding the pathophysiological mechanisms of the disease, is a significant problem for clinical practice.

Due to the steady increase in the burden of HFpEF, especially in women, it is an important task to search for new markers and early predictors associated with the development of this disease. This area of scientific activity has become especially popular in recent years in both world and domestic cardiology. The leading causes of the development of HFpEF are old age, obesity, coronary heart disease and pulmonary hypertension. A significant association has also been established with such markers as female gender, diabetes mellitus (DM), chronic kidney disease (CKD), alcohol abuse, arterial hypertension, smoking and others. Important issue now is the study of the association of pregnancy factors and its complications with the development of various forms of HF in both early and long-term periods. It is known that significant changes in a woman's body during pregnancy contribute to the development of important structural and hemodynamic changes in the cardiovascular system, which, in the absence of predisposing adverse factors, are in most cases reversible. Unfortunately, pathology detected during pregnancy is also often a trigger factor for the formation of structural remodeling of the heart and blood vessels, which can lead to the development of HF in the long term after pregnancy.

Despite the presence of large foreign studies reflecting the high incidence of various forms of chronic non-communicable diseases in women with adverse in the gestational period, the relationship of adverse pregnancy outcomes (APOs) with the development of long-term cardiac pathology, in particular, HFpEF, has not been sufficiently studied. Moreover, approaches to the diagnosis of HFpEF vary significantly, there are often no diagnostic protocols in the studies. In such works, a universal approach is more frequently used without dividing patients into phenotypes, depending on age and comorbidity ("one-size-fits-all approach"), which is critically important in assessing such a heterogeneous disease. The above factors make the interpretation of the data and conclusions ambiguous.

To date, the issue of the association of adverse pregnancy factors with the development of HFpEF in the long-term period is unsolved. It is particularly interesting to study the younger phenotype of patients due to the greater detectability of HFpEF in this group of individuals in Russia compared with Western countries. Studying the nature of this relationship will expand understanding of the role of different APOs in the development of structural and functional changes of the heart in a woman's future.

ELIGIBILITY:
Inclusion Criteria:

* All patients who administer to the Federal State Budgetary Institution National Medical Research Center for Therapy and Preventive Medicine, who are undergoing echocardiography for medical reasons
* Pregnancy >20 weeks in the anamnesis
* Signed informed consent to participate in the study

Exclusion Criteria:

* Refusal to sign an informed consent to participate in a clinical trial and to process personal data
* Detection of left ventricle ejection fraction < 50% according to Echocardiography data

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Generic Moscow population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
HFpEF incidence | on enrollment
  Heart Failure with Preserved Ejection Fraction will be assessed with the transthoracic echocardiography based on the criteria of American Heart Association guidelines, where left ventricle ejection fraction > 50%.
APOs incidence | on enrollment
  Adverse pregnancy outcomes will be determined by means of questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Olga Dzhioeva, MD, PhD, Study Director — National Medical Research Center for Therapy and Preventive Medicine
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No